CLINICAL TRIAL: NCT04124146
Title: Long-term Evolution of Patients Suffering From Lumbar Canal Stenosis and Supported by Minimally Invasive Surgery
Brief Title: Long-term Evolution of Patients Suffering From Lumbar Canal Stenosis and Supported by Minimally Invasive Surgery: SUIVISTENO
Acronym: SUIVISTENO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Medico-Chirurgicale et Obstetrique Cote d'Opale (Network)
Responsible Party: Sponsor
Other Study IDs: SUIVISTENO
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Surgery more than 10 years: Patients with surgery for spinal lumbar stenosis between 2006 and 2008 will be purposed to participate to the study.
  Interventions: Radiation: MRI for some patients according functionnal tests results

INTERVENTIONS:
Radiation: MRI for some patients according functionnal tests results — Depending on the results obtained on the evaluation criteria, additional examinations could be prescribed (imaging) for subjects with an unsatisfactory functional score. There is therefore a potential change in the usual care.

SUMMARY:
describe the functional evolution of patients at more than 10 years post intervention.

describe the evolution of pain, satisfaction, quality of life of patients to more than 5 years pot intervention.

DETAILED DESCRIPTION:
Stenosis of the lumbar canal is a degenerative disorder, occurring most often in the elderly or middle aged, after 50 years. It most often results from the combination of 2 pathologies: the congenital narrowness of the lumbar canal is decompensated over time by the anatomical reorganizations generated by osteoarthritis. It is classically manifested by pain in the lower limbs, occurring almost exclusively in walking or in case of prolonged standing. This postural and dynamic character of the symptomatology is very characteristic of this pathology. The levels most often involved are L4 / L5 and L3 / L4. But, in case of extensive stenosis, other levels may be involved (L2 / L3, L5S1 or even L1 / L2).

Surgical treatment is obviously indicated from the outset in emergency situations or in cases of severe functional disability. It is most often proposed in case of failure of a complete and well-conducted medical treatment. In practice, in cases of tight canal stenosis, only a surgical operation can relieve the patient of pain and recover a normal walk.

A minimal invasive technique: lumbar recalibration, which consists of decompression of the roots of the horse's tail under a microscope without fusion, without arthrodesis, provides a short-term functional benefit, even when Grade 1 spondylisthesis exists. The interest of this technique for the patient is twofold: first aesthetic because the incision is much smaller than in the classical technique and becomes almost invisible after a few months; then and above all it is functional because, by preserving the paravertebral muscles that it allows, this procedure is less painful and allows a lift the same day and an earlier recovery activities.

Very few scientific publications compare different surgical techniques, and even fewer results are available on the long-term future of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated within the institution between 2006 and 2008
* Major patient (18 years old or over).
* Francophone.
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or lactating women according to article L1121-5 of the CSP.
* Vulnerable persons according to article L1121-6 of the CSP.
* Major persons placed under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been cared for at the institution between 2006 and 2008 (cohort) will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
sub-functional score | Month 1
  items VIII to XII of the Swiss Spinal Stenosis questionnaire (French version).

SECONDARY OUTCOMES:
Swiss Spinal Stenosis questionnaire (French version) | Month 1
  under scores symptoms and satisfaction of the Swiss Spinal Stenosis questionnaire (French version)
EQ5D questionnaire | Month 1
  under scores satisfaction of the EQ5D questionnaire
Scale of assessment of lower back pain, leg and when walking | Month 1
  VAS scale scores

IPD SHARING:
Plan to Share IPD: No
The source documents are the original documents, the data and the files, from which the data concerning the research participants are reported in the observation notebook. Excel file that can be opened from a password